CLINICAL TRIAL: NCT01234610
Title: Exercise Therapy for Abdominal Aortic Aneurysm Disease: a Feasibility Study
Brief Title: Feasibility Study of Exercise Training for Abdominal Aortic Aneurysm Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH15455
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Aortic Aneurysm, Abdominal; Aneurysm; Aortic Disease; Vascular Disease; Cardiovascular Disease
Keywords: Exercise; Aortic aneurysm; Feasibility; Vascular disease
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm; Aortic Diseases; Vascular Diseases; Cardiovascular Diseases; Motor Activity; Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): Exercise
  Interventions: Behavioral: Supervised exercise training
- Control (No Intervention): No exercise

INTERVENTIONS:
Behavioral: Supervised exercise training — Patients will be asked to attend three exercise sessions per week for 12 weeks. They will exercise in groups of up to four per session and they will be supervised by an experienced exercise physiologist. Each session will comprise 5 to 10 min warm-up period (involving very light aerobic exercise and a range of gentle movements), 30 min of light-to-moderate intensity aerobic exercise (cycle-ergometry and or treadmill-walking), and a 5 to 10 min cool-down period involving low-intensity aerobic exercise and gentle stretching. The intensity of the aerobic exercise will be individualised and will be progressed gradually (if appropriate) during the course of the study.
  Arms: Exercise

SUMMARY:
An abdominal aortic aneurysm (AAA) is a weakened and enlarged area in the abdominal aorta, which is a large blood vessel in the abdomen. Large AAAs (>55 mm diameter) carry a high risk of rupture, a surgical emergency that often leads to death due to severe internal bleeding. It has been suggested that regular exercise training might limit the rate at which AAAs develop. However, little is known about the safety and effectiveness of exercise training in these patients. This pilot study will examine the feasibility of supervised aerobic exercise training for patients with small AAAs (30 to 49 mm diameter). The investigators hypothesize that exercise training will be safe and useful for patients with small AAAs.

DETAILED DESCRIPTION:
Abdominal aortic aneurysm (AAA) disease is a potentially lethal health problem of older adults. New screening initiatives will identify many individuals with small (30 to 49 mm) AAAs for which there are currently no treatment options. Regular aerobic exercise might retard AAA disease progression, but the feasibility and acceptability of aerobic exercise in patients with AAA disease has yet to be established. This pilot study will examine the feasibility of supervised aerobic exercise and exercise advice-only in patients with small AAAs. A total of 60 volunteers will be recruited and randomly allocated to one of the two groups. Patients in the supervised exercise programme will be offered three supervised cycle ergometry/treadmill-walking sessions for a period of 12 weeks. The feasibility of each intervention will be assessed in terms of recruitment and compliance, attrition, changes in cardiopulmonary fitness and objective measures of free-living physical activity. Changes in aneurysm size and blood markers associated with disease progression will also be monitored and the impact of the interventions on health-related quality of life assessed using a questionnaire. Outcomes will be assessed at baseline and 12 weeks. We will also conduct focus groups at the end of the trial to obtain qualitative feedback from patients. The results of this study will inform the design of a multi-centre randomised controlled trial with longer-term follow-up of clinical end-points.

ELIGIBILITY:
Inclusion Criteria:

* Men or women identified as having a stable 30 to 49 mm asymptomatic, infra-renal AAA, measured using high-resolution B-mode ultrasonography
* Ability to undertake exercise testing and training

Exclusion Criteria:

* Patients with large (>50 mm)/symptomatic AAAs
* Patients with contraindications to exercise testing/training (e.g. severe hypertension, unstable metabolic/cardiopulmonary conditions, musculoskeletal injuries etc…)
* Patients who are unable to travel to the testing and training facility at Sheffield Hallam University
* Patients who are already participating in regular exercise
* Patients with a mental impairment that would render consent unethical or would make compliance difficult (e.g. dementia or Alzheimer's)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Feasibility | 12 weeks
  We will monitor how feasible it is to recruit, test and train patients with small AAAs

SECONDARY OUTCOMES:
Cardiopulmonary fitness | 12 weeks
  Peak oxygen uptake and ventilatory threshold assessed during an incremental-load cycling test
Quality of life | 12 weeks
  Health-related quality of life assessed using the MOS SF-36 v2 questionaire
Aneurysm size | 12 weeks
  Aneurysm size as measured using B-mode ultrasound
Blood biomarker of disease progression | 12 weeks
  Fasting blood samples will be taken to assess changes in hs-CRP
Blood biomarker of disease progression | 12 weeks
  Fasting blood samples will be taken to assess changes in MMP-9

CONTACTS AND LOCATIONS:
Overall Officials: Shah Nawaz, MD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust; Garry A Tew, PhD, Principal Investigator — Sheffield Hallam University
Locations (2):
- United Kingdom (2):
  - Sheffield Hallam University, Sheffield, South Yorkshire
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire